CLINICAL TRIAL: NCT05655273
Title: Prograf/Envarsus Conversion Study in Liver Transplant Recipients to Improve Side Effects, Adherence and Quality of Life: a Single-centre Randomized Controlled Trial
Brief Title: Conversion of Maintenance Prograf to Envarsus in Liver Transplant Recipients
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Paladin Labs Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-5210
Record Dates: First submitted 2022-11-22; First posted 2022-12-19 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Liver Transplant Rejection; Immune System Suppression
Keywords: liver transplant; tacrolimus toxicity; drug conversion; tacrolimus; prograf; envarsus
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: conversion v. control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Post-liver transplant patients receiving Prograf (Active Comparator)
  Interventions: Drug: Prograf
- Post-liver transplant patients receiving Envarsus (Active Comparator)
  Interventions: Drug: Envarsus

INTERVENTIONS:
Drug: Prograf — Participants randomized to the Prograf (control) arm will continue with their current twice daily dosing of Prograf.
  Arms: Post-liver transplant patients receiving Prograf
Drug: Envarsus — Participants randomized to Envarsus arm will have their current daily dose of Prograf converted to once-daily Envarsus dose according to the following ratio: 0.7 x the current daily Prograf dose. Envarsus is available in 3 dose strengths- 0.75mg, 1.0mg, and 4.0mg. The actual dose of Envarsus will be rounded to an amount that can be administered using the above tablet strengths.
  Arms: Post-liver transplant patients receiving Envarsus

SUMMARY:
Prograf and Envarsus are two different formulations of Tacrolimus which is used as an immunosuppressant in liver transplant (LT) patients. Prograf is currently used as part of the standard immunosuppression regimen for LT recipients at UHN. This study will compare the use of Prograf and Envarsus and their effects on liver and renal function, trough tacrolimus levels, drug-related adverse effects, and patient adherence. Trial design is a pilot randomized trial. The study aims to recruit 40 patients from UHN's LT program and they will be randomized 1:1 to either stay on their current dose of Prograf or be converted to a once-daily equivalent dose of Envarsus. Both groups of patients will be followed for 48 weeks. This study will compare the change from baseline to week 48 in liver and renal function, tacrolimus-related side effects and patient reported outcomes between the two study groups.

DETAILED DESCRIPTION:
Tacrolimus (Prograf ©) has become part of the standard of care for patients receiving solid organ transplants and is part of the immunosuppressive protocol (along with prednisone and mycophenolate mofetil [CellCept ©]) used by liver transplant recipients at University Health Network (UHN). Tacrolimus is associated with several toxicities including renal injury, tremor, pancreatic islet β-cell injury (leading to diabetes) and hyperlipidemia. As a result of these potential toxicities, careful therapeutic drug monitoring of tacrolimus is a key component of post-transplant management. Tacrolimus trough levels are known to correlate with total tacrolimus exposure, as shown from formal pharmacokinetic assessments. Accordingly, trough serum concentrations of tacrolimus are measured routinely in all recipients and are used to guide dosing. The Prograf formulation of tacrolimus has a short serum half-life and must be dosed twice daily to maintain therapeutic serum concentrations. Further, Prograf administration results in a high peak tacrolimus level. Peak tacrolimus levels have been shown to correlate with toxicity; thus, avoidance of high peaks may be desirable to minimize tacrolimus toxicity.

Envarsus is an extended-release formulation of tacrolimus that provides similar drug exposure to tacrolimus at a 30% lower dose but with a once daily dosing regimen. Envarsus dosing also results in a lower peak tacrolimus level compared to Prograf. In this way, it is hoped that Envarsus may provide similar therapeutic efficacy as Prograf but with fewer adverse effects. In addition, the simpler dosing regimen is expected to enhance patient adherence and quality of life.

The present study is aimed at evaluating the impact of a switch from Prograf to Envarsus on liver and renal function, trough tacrolimus levels, drug-related adverse effects and adherence. It hypothesizes that once daily Envarsus can be substituted at reduced daily dose for twice daily Prograf in stable liver transplant recipients without clinically meaningful changes in liver allograft function while reducing tacrolimus side effects, reducing cumulative daily dose of the drug and increasing adherence to treatment and quality of life.The results of this study have the potential to change current practice. Trial design is a pilot randomized trial. The study aims to recruit 40 patients from UHN's LT program and they will be randomized 1:1 to either stay on their current dose of Prograf or be converted to a once-daily equivalent dose of Envarsus. Both groups of patients will be followed for 48 weeks. This study will compare the change from baseline to week 48 in liver and renal function, tacrolimus-related side effects and patient reported outcomes between the two study groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years) prevalent liver transplant recipient
* >12 months after liver transplant
* Prograf-based maintenance immunosuppression with targeted tacrolimus trough level of 5-10 ug/L
* Stable liver allograft function (defined as ASL & ALT <30, Bilirubin <20 & ALP<150 at baseline visit or within 4 weeks of baseline visit)
* Stable renal function (creatinine < 180 µmol/l and eGFR > 40 ml/min) at baseline visit (or within 4 weeks of baseline visit)
* No episode of acute rejection within 6 months of baseline visit
* Elevated creatinine (defined as >ULN) OR Significant symptoms (by patient self-report) potentially associated with tacrolimus (eg. tremor, difficulty to concentrate, insomnia) OR difficulty to adhere to a twice daily regimen

Exclusion Criteria:

* Multiorgan transplant;
* severe intercurrent illness;
* severe cognitive impairment (all as determined by clinical team);
* unwilling to consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in AST levels | Baseline to week 12
Change in ALT levels | Baseline to week 12
Change in ALP levels | Baseline to week 12
Change in Bilirubin blood levels | Baseline to week 12
Change in tacrolimus trough levels | Baseline to week 12
Change in overall daily dose of tacrolimus | Baseline to week 12

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure | Baseline to week 24 and week 48
Change in Diastolic Blood Pressure | Baseline to week 24 and week 48
Change in Renal function (eGFR) | Baseline to week 24 and week 48
Change in tremor severity (for subset of patients who report significant tremor at baseline) | Baseline to week 24 and week 48
Change in glycemic control (HbA1c) | Baseline to week 24 and week 48
Change in lipid profile | Baseline to week 24 and baseline to week 48
Change in Patient-Reported Outcomes Measurement Information Systems' Pain Interference Bank 2.0 | Baseline to Week 48 (inclusive)
Change in Patient-Reported Outcomes Measurement Information Systems' (PROMIS) Sleep Disturbance Bank 1.0 | Baseline to Week 48 (inclusive)
Change in Patient-Reported Outcomes Measurement Information Systems' (PROMIS) Anxiety Bank 1.0 | Baseline to Week 48 (inclusive)
Change in Patient-Reported Outcomes Measurement Information Systems' (PROMIS) Depression Bank 1.0 | Baseline to Week 48 (inclusive)
Change in Patient-Reported Outcomes Measurement Information Systems' (PROMIS) Global Health Scale version 1.2 | Baseline to Week 48 (inclusive)
Change in Patient-Reported Outcomes Measurement Information Systems' (PROMIS) Fatigue bank 1.0 | Baseline to Week 48 (inclusive)
Change in Patient-Reported Outcomes Measurement Information Systems' (PROMIS) Ability to Participate in Social Roles and Activities | Baseline to Week 48 (inclusive)

CONTACTS AND LOCATIONS:
Overall Officials: Nazia Selzner, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No